CLINICAL TRIAL: NCT04144920
Title: Evaluating the Acute Glycemic Response to Different Strategies of Breaking Up Sedentary Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Matthew P Buman, PhD, Associate Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00008450
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Pre Diabetes; Postprandial Hyperglycemia
Keywords: Interrupting sitting; Continuous glucose monitroing; Pattern of sitting breaks
MeSH Terms: conditions — Glucose Intolerance; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: The study design is a crossover randomized trial with three conditions: (i) uninterrupted sitting, (ii) high-frequency and low duration (HFLD) standing breaks, and (iii) low-frequency and high duration (LFHD) standing breaks. We utilized a balanced and uniform with 6 randomization blocks (ABC, ACB, BAC,BCA, CAB, CBA) design.
Who Masked: Participant
Masking Description: Participants were blinded on what protocol they will be performing until after their first standardized meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Block 1 (Other): Participants in this arm performed the conditions in this order: CS, HFLD, LFHD
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks
- Block 2 (Other): Participants in this arm performed the conditions in this order: CS, LFHD, HFLD
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks
- Block 3 (Other): Participants in this arm performed the conditions in this order: HFLD, CS, LFHD
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks
- Block 4 (Other): Participants in this arm performed the conditions in this order: HFLD, LFHD, CS
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks
- Block 5 (Other): Participants in this arm performed the conditions in this order: LFHD, CS, HFLD
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks
- Block 6 (Other): Participants in this arm performed the conditions in this order: LFHD, HFLD, CS
  Interventions: Behavioral: CS: Continuous sitting; Behavioral: HFLD: HIgh frequency, low duration standing breaks; Behavioral: LFHD: Low frequency, high duration standing breaks

INTERVENTIONS:
Behavioral: CS: Continuous sitting — Participants were asked to sit continuously throughout the duration of the lab visit.
Behavioral: HFLD: HIgh frequency, low duration standing breaks — Participants were asked to interrupt their sitting time every 15 minutes using 2.5-minute standing breaks.
Behavioral: LFHD: Low frequency, high duration standing breaks — Participants were asked to interrupt their sitting time every 60 minutes using 10-minute standing breaks.

SUMMARY:
This study aims to determine the most effective strategy of reducing sedentary behavior to improve health. Specifically, we aim to answer the following questions: (a) To determine if there is a significant difference in acute post-prandial glucose response between continuous sitting and two intermittent standing regimes (high frequency, low duration breaks (HFLD) and low frequency, high duration breaks (LFHD)). We hypothesize that intermittent standing (combined HFLD breaks and LFHD breaks regimes) will result in lower overall acute post-prandial glucose compared to continuous sitting. (b) To determine if there is a significant difference in acute post-prandial glucose response between two strategies to reduce sitting with standing (HFLD standing breaks vs. LFHD standing breaks). We hypothesize that the HFLD breaks condition will elicit lower acute post-prandial glucose level compared to the LFHD breaks condition. All eligible participants will be consented and subjected to all three study conditions: (i) Uninterrupted sitting, (ii) HFLD breaks, and (iii) LFHD breaks. The order at which participants were subjected to these conditions will be randomly determined and each condition were performed a week apart. Standardized meals (breakfast and lunch) will be provided during each lab visit and participants will be then be asked to perform their usual work activity using a sit-stand workstation in the lab. Depending on their assigned condition, the participants will be prompted to stand or sit for a given period of time. A continuous glucose monitor will be used to measure glucose response to the intervention while an activPAL device will be used to make sure that participants are compliant with the study protocol.

DETAILED DESCRIPTION:
Most studies that explored the health benefits of interrupting sitting time focused on using different modalities (i.e., comparing walking vs standing breaks). However, experimental studies that directly compare patterns of interrupting sitting time through standing only are needed to advance the field. This study aimed to (i) determine if there is a difference in glucose response between continuous sitting (CS) and two intermittent standing regimes (high frequency, low duration breaks (HFLD) and low frequency, high duration breaks (LFHD)) and (ii) to determine if there is a difference in glucose response between the two strategies (HFLD vs. LFHD).

A. Study Participants and Recruitment The target participants were sedentary office employees with impaired fasting glucose level. Participants were recruited through a study flyer via various recruitment channels (i.e., ASU faculty website, social media, word of mouth). The study flyer contains a link to a Qualtrics survey to pre-screen interested participants. All eligible participants will be scheduled for a 30-minute screening visit to assess fasting glucose level. A total of 12 sedentary and inactive employees (indicated by >6 hrs of workplace sedentary time assessed by the activPAL device during a one-week screening period) will be enrolled to participate in a fully randomized crossover trial.

B. Study Design The study design is a crossover randomized trial with three conditions: (i) uninterrupted sitting, (ii) high-frequency and low duration (HFLD) standing breaks, and (iii) low-frequency and high duration (LFHD) standing breaks. In the interrupted sitting conditions (i.e., HFLD and LFHD), total sitting and standing time were designed to be equal in both groups. The only difference between the two conditions was on the pattern to accumulate sitting time. A common threshold for prolonged sitting time in epidemiological studies of sedentary behavior is 30 minutes of continuous sitting. In the HFLD condition, we will use half of this threshold and ask participants to interrupt their sitting time every 15 minutes using a 2.5-minute standing break. In contrast, participants will perform twice this threshold in the LFHD standing breaks where they will complete a 10-minute standing break every hour of sitting.

All possible sequence of condition were determined and organized into blocks (a total of six blocks). Each eligible participant will be randomly assigned to a block to determine the sequence that they would perform the conditions. The randomization process will involve a separate research staff preparing 40 sealed envelope that contains a block number randomly determined using a computer-generated random sequence. These envelopes will be kept in a secure cabinet by another research staff not directly involved in the project. Each participant will be blinded to the condition that they are going to perform during the visit until after their first standardized meal.

Participants will be invited to three 450-minute (7.5-hour) laboratory visits where they will be provided with a private room, a sit-stand workstation, and a desktop computer. During each laboratory visit, participants will perform their usual desk-based work activities. All visits will be scheduled one week apart. Participants will be instructed to fast overnight, and standardized breakfast and lunch meals will also be provided to control for any dietary effects on glucose level. In addition, each participant will be instructed to avoid any moderate-vigorous physical activities for at least two days and smoking cigarettes and consuming alcoholic beverages at least three days prior to each visit. Upon arrival to the lab for their first visit, participants will complete a dietary log of their last meal the previous day. They will then be instructed to replicate this meal the night prior to each visit.

C. Outcome Measures Continuous Glucose Monitors. A day prior to the first visit, participants will be fitted with a Freestyle Libre Pro (Abbott Laboratories, Chicago, IL) continuous glucose monitor by a trained researcher. The sensor will be attached to the back part of the participant's non-dominant arm and programmed to measure interstitial glucose at 15-minute intervals. The device is designed to be worn continuously for 14 days and is waterproof, lightweight (roughly the size of a quarter) and minimally obtrusive. The sensors will be attached using proper aseptic procedures and in accordance with the manufacturer's instructions. Lastly, each participant will be given instructions on how to care for the device.

At the end of the last visit, data from each sensor will be acquired using the Libre Pro reader and uploaded to an online patient repository (LibreView). Data will then be processed, and 15-minute epoch data will be downloaded into a local secure drive for further processing. Continuous glucose data corresponding to each visit date and time will be isolated using the paper logs and inspected for completeness and quality of data. Files with less than 80% of valid observation will be excluded from the succeeding analyses. Glucose incremental area under the curve (iAUC) will be calculated using the trapezoidal method along with other metrics for variability (i.e., MAGE: mean amplitude of glycemic excursions).

activPAL Device. Objective measures of sitting, standing and moving time will derived from the activPAL micro accelerometer worn on the midline of the right thigh. Participants will wear the device on two occasions: (i) for 7 consecutive days during the baseline period and (ii) for 14 consecutive days during the study. The validity and reliability of the activPAL in measuring sedentary and physical activity behaviors has been previously reported. Collected data will be processed into events of sitting, standing, or moving (i.e., stepping) using the activPAL software version 7.2.32 (PAL Technologies Ltd, Scotland, UK).

Standard Meals. Standardized meals (breakfast and lunch) will be provided in each lab visit to control for any dietary influence. Each meal are designed to provide 33% of the participant's total daily caloric needs following a typical American diet (50-60% carbohydrates, 25-35% fat, and 10-20% protein). Basal metabolic rate will be calculated for each particiapnt using Schofield's equation using a 1.5 activity factor. After calculating the required caloric content of each meal, a meal with the closest caloric value will be chosen from a list of pre-determined meal plan. A typical breakfast will be composed of a croissant, ham, cheddar cheese, cereals with milk, fruit cup, and orange juice while lunch items consisted of a ciabatta ham and cheese sandwich and orange juice. The same meal will be provided during all follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

(i) ages 35-65 years, (ii) sedentary work habits, (iii) presence of impaired fasting glucose (fasting glucose level of 100-125 mg/dL), (iv) willing to engage in three 7.5 hour lab visit, (v) willing to wear the activPAL and continuous glucose monitor, (vii) current sit-stand workstation owner, and (viii) BMI 25-45 kg/m2

Exclusion Criteria:

(i) chronic mobility limitations, such as moderate-to-severe arthritis, (ii) psychiatric disorders, (iii) cardiometabolic abnormality, (iv) food allergy/restriction, (v) BMI>45 kg/m2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose incremental area under the curve (iAUC) | post breakfast (3.5 hrs), post lunch (3.5 hrs), and total lab time (7 hrs)
  iAUC will be calculated using the trapezoidal method.
Mean postprandial glucose | post breakfast (3.5 hrs), post lunch (3.5 hrs), and total lab time (7 hrs)
Glucose variability (mean amplitude glycemic excursions) | total lab time (7 hrs)

SECONDARY OUTCOMES:
Physical and Emotional feeling states | total lab time (7 hrs)
  Self-report (via EMA) measures of fatigue, stress, busyness, hunger, and affective states

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided